CLINICAL TRIAL: NCT06661902
Title: BURN Study: Buffered Lidocaine in Reducing Pain From Prostate Biopsy
Brief Title: Buffered Lidocaine for Reducing Pain in Patients Undergoing Prostate Biopsy, BURN Trial
Acronym: BURN
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: RG1125023; STUDY00021446 (Other: Fred Hutch/University of Washington Cancer Consortium); NCI-2024-10011 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2024-10-25; First posted 2024-10-28 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; prostate biopsy; transperineal biopsy; transrectal biopsy; MRI fusion biopsy; buffered lidocaine; sodium bicarbonate; Local anesthesia; lidocaine
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Lidocaine; Sodium Bicarbonate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The Investigational Drug Services team will be unblinded to the patient's randomization status. During statistical analysis of the data, the statistician will be concealed to the randomization allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (lidocaine) (Active Comparator): Patients receive SOC lidocaine via injection during SOC prostate biopsy on study.
  Interventions: Drug: Lidocaine; Procedure: Biopsy of Prostate; Other: Questionnaire Administration
- Arm B (buffered lidocaine) (Experimental): Patients receive buffered lidocaine via injection during SOC prostate biopsy on study. (1% Lidocaine + 8.4% Sodium Bicarbonate, in a 3:1 ratio)
  Interventions: Drug: Buffered Lidocaine (1% Lidocaine + 8.4% Sodium Bicarbonate, in a 3:1 ratio); Procedure: Biopsy of Prostate; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Buffered Lidocaine (1% Lidocaine + 8.4% Sodium Bicarbonate, in a 3:1 ratio) — Given via injection
  Arms: Arm B (buffered lidocaine)
Drug: Lidocaine — Given via injection
  Arms: Arm A (lidocaine)
Procedure: Biopsy of Prostate — Undergo SOC prostate biopsy
  Other Names: Prostate Biopsy
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase I/II trial examines if buffered lidocaine reduces the pain that patients may experience during prostate biopsy. Prostate biopsies are typically performed awake, in the office, with only local anesthetic. As a result, many patients note considerable pain during these procedures. Local anesthetics such as lidocaine are typically acidic, which is thought to cause pain and burning during infiltration (injection). As a result, buffered local anesthetic has become the standard of care (SOC) in multiple specialties using awake local anesthetic. However, it has not been explored during prostate biopsies. Adminstering buffered lidocaine may reduce pain in patients undergoing prostate biopsy.

DETAILED DESCRIPTION:
OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A: Patients receive SOC lidocaine via injection during SOC prostate biopsy on study.

ARM B: Patients receive buffered lidocaine via injection during SOC prostate biopsy on study.

After completion of study intervention, patients are followed up 1-2 days post-biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* 18 years old or older
* Patients with prostates
* Those with and without a prior diagnosis of prostate cancer
* Recommended to undergo a prostate biopsy in the urology clinic. Only patients that have been scheduled for a biopsy (for clinical purposes) will be enrolled. May include all of the following types of prostate biopsies:

  * Transperineal or transrectal
  * Systematic or targeted/fusion biopsy
  * 12 core biopsy or > 12cores
  * Biopsy naïve or prior biopsy

Exclusion Criteria:

* Anorectal pathology precluding placement of a transrectal ultrasound
* Diagnosis of chronic prostatitis, interstitial cystitis, pelvic pain syndrome
* Concomitant chronic pain condition
* Neurological condition affecting pain or sensorium (ex. spinal cord injury, stroke, multiple sclerosis, etc.)
* Prostate biopsy performed with any anesthesia other than local anesthetic (monitored anesthesia care, general anesthesia)
* Prostate biopsy completed in the operating room
* Patients who ultimately require additional local anesthetic beyond what is allotted in the study intervention
* Patients taking anxiolytics in the 6-hours prior to the biopsy
* Those with a known hypersensitivity, allergic reaction, or contraindication to using sodium bicarbonate. This includes patients who are receiving diuretics known to produce a hypochloremic alkalosis

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2025-01-09 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Pain of Local Anesthetic Injection | Within 20 seconds of completing the injection of all local anesthetic
  Pain associated with the injection of local anesthetic, assessed by a written questionnaire (Visual Analogue Scale, 0 [least] to 10 [worst pain]).

SECONDARY OUTCOMES:
Pain of the Prostate Biopsy | Within 10 minutes of completing the prostate biopsy, and on post-operative day 1
  Pain associated with the biopsies of the prostate, assessed by a questionnaire (Visual Analogue Scale, 0 [least] to 10 [worst pain]).
Willingness to perform another prostate biopsy in the future, if medically necessary | Within 10 minutes of completing the prostate biopsy, and on post-operative day 1
  Assessed by a questionnaire (Visual Analogue Scale, 0 [least likely] to 10 [most likely])
Incidence of adverse events | Post-operative day 1
  Will be assessed by patient self-report using an electronic written questionnaire. Will be assessed for inability to urinate, bleeding, allergic reaction, fever, or fatigue, or significant chills, or nausea/vomiting.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Zhu, DO, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No
This is a single center, investigator initiated trial.